CLINICAL TRIAL: NCT01097252
Title: Randomized Trial of Concurrent Chemoradiation With Weekly Versus Three-week Cisplatin in Patients With Advanced Cervical Cancer
Brief Title: Weekly Versus Three-week Chemoradiation in Patients With Advanced Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Cancer Center Hospital (Other)
Responsible Party: Principal Investigator, Sang-Young Ryu, Chair of Cerivcal/Ovarian Cancer Center, Korea Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCCH GY 1005
Record Dates: First submitted 2010-03-29; First posted 2010-04-01 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Cervical Cancers
Keywords: Cervical Neoplasm; chemoradiation; compliance; toxicity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Patient Compliance | interventions — Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- weekly cisplatin (Active Comparator): Weekly cisplatin 40mg/m2 during radiation therapy
  Interventions: Radiation: radiation; Drug: weekly cisplatin
- tri-weekly cisplatin (Experimental): cisplatin 75mg/m2 three cycles, every 3 weeks
  Interventions: Radiation: radiation; Drug: tri-weekly cisplatin

INTERVENTIONS:
Radiation: radiation — radiation with cisplatin 40mg/m2, 6 cycles, every week
Drug: weekly cisplatin — weekly cisplatin 40mg/m2, 6 cycles
  Other Names: Cisplatin
  Arms: weekly cisplatin
Drug: tri-weekly cisplatin — cisplatin 75mg/m2, 3cycles, every 3 weeks
  Other Names: Cisplatin
  Arms: tri-weekly cisplatin

SUMMARY:
Three weekly cisplatin based chemoradiation is to be compared the compliance, toxicity, and response rates with the weekly cisplatin based chemoradiation in the treatment of locoregionally advanced cervical cancers.

DETAILED DESCRIPTION:
This study is to compare the compliance, toxicity, response and survival rate between concurrent chemoradiation with weekly cisplatin 40mg/m2 and three-week cisplatin 75mg/m2 in patients with advanced cervical cancer. Patients with primary untreated invasive squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix from stage IIB to IVA were enrolled. Patients with histologically proven locoregionally advanced cervical cancer will be randomized into two treatment arm; Arm I, concurrent chemoradiation with weekly cisplatin 40mg/m2 for six times; Arm II, concurrent chemoradiation with three-week cisplatin 75mg/m2 for three times. The compliance and toxicity during the chemoradiation is the primary endpoint. Response rate and the overall survival will be analyzed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cervical cancer
* Squamous, Adenosquamous, Adeno carcinoma cell type
* International Federation of Gynecologic Oncology (FIGO) stage IIB - IVA
* Gynecologic Oncology Group (GOG) performance status 0 - 2

Exclusion Criteria:

* Previous history of chemotherapy or radiation
* History of other cancer
* Hypersensitivity to platinum agents
* Pregnancy
* Serious medical disease

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2002-01; Primary Completion 2004-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
compliance | 3 month
  1. Percentage of completed cycles of scheduled chemotherapy in each arm
  2. Percentage of grade III and IV toxicity
  3. Delayed radiation time due to toxicity

SECONDARY OUTCOMES:
survival | 5 years
  1. 5 year progression free survival
  2. 5 year survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Young Ryu, MD, Principal Investigator — Korea Institute of Radiological & Medical Sciences
Locations (1):
- Korea Institute of Radiological & Medical Sciences, Seoul, South Korea

REFERENCES:
- [Result] Ryu SY, Lee WM, Kim K, Park SI, Kim BJ, Kim MH, Choi SC, Cho CK, Nam BH, Lee ED. Randomized clinical trial of weekly vs. triweekly cisplatin-based chemotherapy concurrent with radiotherapy in the treatment of locally advanced cervical cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e577-81. doi: 10.1016/j.ijrobp.2011.05.002. Epub 2011 Aug 11. PMID 21840137